CLINICAL TRIAL: NCT05582174
Title: A Comparison Between a High Dose PPI Intravenous Infusion and Oral Acid Pump Inhibitors After Endoscopic Haemostasis to Bleeding Peptic Ulcers
Brief Title: PPI Infusion Versus Oral Acid Pump Inhibitors for Bleeding Peptic Ulcers
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, MD, professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPI vs VPZ study
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Upper GI Bleeding; Proton Pump Inhibitors
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole

STUDY DESIGN:
Who Masked: Investigator
Masking Description: random sequence was investigator-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PPI infusion (Active Comparator): esomeprazole 80mg iv bolus followed by 8mg per hour for 72 hours
  Interventions: Drug: esomeprazole
- Vonoprazan (Experimental): Vonoprazan 40 mg bid orally for 72 hours, and from day 4-30 VPZ 20 mg daily
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan 40 mg bid orally for 72 hours, and from day 4-30 VPZ 20 mg daily
  Other Names: Takecab
  Arms: Vonoprazan
Drug: esomeprazole — A high dose PPI infusion (esomeprazole 80mg iv bolus followed by 8mg per hour for 72 hours), and frorm day 4-30 oral esomeprazole daily
  Other Names: nexium
  Arms: PPI infusion

SUMMARY:
Vonoprazan (VPZ), an oral potassium-competitive acid blocker (P-CAB) has emerged as an alternative potent acid-suppressant.It has a faster onset of action in 1 day (3-5 days in PPI), and is more stable in acidic condition than PPI. While many studies compared Vonoprazan against PPI in the treatment of reflux oesophagitis, H. Pylori eradication, and gastric ulcers; thus far, there is a paucity of data on use of Vonoprazan on bleeding peptic ulcers.

We perform a multicenter randomized controlled trial (RCT) to compare the efficacy of oral Vonoprazan against standard high dose PPI therapy in bleeding peptic ulcers that had received successful endoscopic haemostasis We hypothesize that in patients with bleeding peptic ulcers, the use of acid pump inhibitors Vonoprazan would not be inferior to standard treatment of a bolus plus high dose PPI intravenous infusion at preventing recurrent bleeding after endoscopic haemostasis.

DETAILED DESCRIPTION:
Upper gastrointestinal bleeding (UGIB) remains an important medical emergency. While the annual incidence having decreased from about 100/100,000 adults in 1990s to 61-78/100,000 persons in 2009-2012 , 30-day mortality remains up to 11% . Despite advancement in various endoscopic haemostatic technology, peri-endoscopic management remains paramount to satisfactory outcome in acute non-variceal gastrointestinal bleeding (NVGIB), especially for peptic ulcer bleeding. Indeed, recurrent bleeding leads to prolonged hospital stay and is an independent risk factor for mortality . Current international guidelines advocate the use of high dose proton pump inhibitors (PPI), as defined as ≥80mg daily for ≥3 days, to be given intermittently or continuously after successful endoscopic haemostatic therapy . It is hypothesized that the lowering of gastric acidity by PPI can facilitate formation and stability of clot, as pepsin-induced clot lysis is inhibited when pH is above 4-5 . Studies including RCTs have shown that PPI therapy markedly reduced further bleeding (RR = 0.43,0.33-0.56), mortality (RR = 0.41, 0.22-0.79) and surgery compared (RR = 0.42, 0.25-0.71) with placebo or no treatment . When compared to other acid suppressants such as H2-blocker (H2B), studies have demonstrated superiority of PPI therapy in reducing rebleeding, but not mortality or need for further intervention . Study has shown PPI infusion can achieve intragastric pH 6 holding time ratio (HTR) for 67.8% over first 24 hour and intragastric pH 4 HTR for 90.5% of the period , while the pH 6 HTR for bolus PPI every 12 hour has been shown to be 49.0% . Despite the apparent difference in effect on intragastric pH, the optimal dose of PPI therapy is still not well defined, with data showing comparable outcome between infusion and intermittent dosing.

In recent years, Vonoprazan (VPZ), an oral potassium-competitive acid blocker (P-CAB) has emerged as an alternative potent acid-suppressant. It was first launched in Japan in February 2015 and has shown satisfactory effect and safety profile in treatment of reflux oesophagitis, H. Pylori eradication, NSAID-associated ulcer, endoscopic submucosal dissection (ESD) induced gastric ulcers and peptic ulcer disease, etc . A RCT has demonstrated non-inferiority of Vonoprazan when compared with lansoprazole in peptic ulcer treatment, while other studies also showed non-inferiority of Vonoprazan to PPI treatment in high risk conditions such as patient on dual-antiplatelet therapy or prevention of bleeding from endoscopic submucosal dissection induced gastric ulcers . It has a faster onset of action in 1 day (3-5 days in PPI), and is more stable in acidic condition than PPI. Studies has demonstrated that Vonoprazan 20 mg once daily achieves 63% pH4 HTR after 24 hours; and the median pH4time (intragastric pH ≥ 4 over 24h after ≥ 5 days of therapy) for Vonoprazan after 7 days of 10, 20, 30, and 40 mg once daily was 60.2%, 85.2%, 90.1%, and 93.2%. . Extrapolating those results to pH4time for PPIs suggests that 10 mg of Vonoprazan once daily is approximately equivalent to 60 mg of omeprazole equivalents (OE), or 40mg of esomeprazole; and 20 mg is equivalent to 60 mg OE bid, or esomeprazole 40 mg bid .

While many studies compared Vonoprazan against PPI in the treatment of reflux oesophagitis, H. Pylori eradication, and gastric ulcers; thus far, there is a paucity of data on use of Vonoprazan on bleeding peptic ulcers. Here, we perform a multicenter randomized controlled trial (RCT) to compare the efficacy of oral Vonoprazan against standard high dose PPI therapy, in the form of high dose intravenous bolus injection (80mg) followed by continuous infusion for 72 hours (8mg/h), in bleeding peptic ulcers that had received successful endoscopic haemostasis. With the hypothesis that 10mg Vonoprazan is approximately equivalent to 40mg of esomeprazole, the total volume of bolus injection and 72 hours infusion of 656mg esomeprazole is approximately equivalent to 164mg Vonoprazan. Therefore, we propose a dose of 40mg every 12hours for 72hours for the treatment of bleeding peptic ulcers. As part of the study, we also investigate the effect of Vonoprazan on intra-gastric pH in this clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* - Patients aged ≥18 years who had undergone oesophagogastroduodenoscopy (OGD) for sign and symptoms of aneamia or upper GI bleeding including haematochezia, melaena or haematemesis, and found to a non-variceal upper GI cause of bleeding (peptic ulcers, dieulafoy's lesions, Mallory Weiss tear with active bleeding or major stigmata of haemorrhage
* Major stigmata of recent haemorrhage includes peptic ulcers with spurting or oozing bleeding (Forrest classification Ia and Ib, respectively) ,with a nonbleeding visible vessel (Forrest classification IIa) or an adherent clot (Forrest classification IIb). For peptic ulcers with an adherent clot (Forrest classification IIb), the clot would be lifted (by irrigation using syringe boluses or water pump device, or manipulation with a snare or alligator etc.) and ulcer base examined to look for underlying vessels. Once the clot is removed, any identified underlying active bleeding or nonbleeding visible vessel should receive endoscopic haemostasis
* Patients who had undergone endoscopic hemostatic treatment (a combination of hemoclipping therapy or contact thermocoagulation using multipolar/bipolar electrocautery probes or haemostatic forceps, with or without preinjection of diluted epinephrine. Endoscopic haemostasis is defined as no evidence of bleeding after irrigation and 3 minutes of observation

Exclusion Criteria:

* No consent
* Patients under the age of 18
* Patients who were pregnant or in lactation
* Hypersensitivity to PPI or Vonoprazan or any component of the formulation
* Patients who were found to have tumour bleeding, oesophageal varices as the cause of the NVGIB
* NVGIB due to post therapeutic endoscopic treatment such as gastric polypectomy, endoscopic mucosal resection, endoscopic submucosal dissection etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-01-03 (Estimated); Study Completion 2026-01-03 (Estimated)

PRIMARY OUTCOMES:
The number of recurrent bleeding | within 30 days after randomization
  The number of recurrent bleeding that occurred after 1st endoscopic hemostasis and confirmed by endoscopy

SECONDARY OUTCOMES:
further treatment for hemostasis | within 30 days after randomization
  the rate of patients that required endoscopic treatment/surgery/embolization for hemostasis
Total Days of hospital stay and intensive unit stay | within 30 days after randomization
  hospital stays and intensive unit stays

CONTACTS AND LOCATIONS:
Overall Officials: Side Liu, PhD, Study Director — Southern Medical University - Southern Hospital
Locations (8):
- China (8):
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Shenzhen Pingshan District People's Hospital, Shenzhen, Guangdong
  - The Second Affiliated Hospital The Chinese University of Hong Kong, Shenzhen & Longgang District People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Yangjiang People's Hospital of Guangdong Medical University, Yangjiang, Guangdong
  - Zhuhai People's Hospital (Zhuhai Hospital Affiliated to Jinan University), Zhuhai, Guangdong
  - Prince of Wales Hospital, Hong Kong, Hong Kong SAR

IPD SHARING:
Plan to Share IPD: No